CLINICAL TRIAL: NCT06787586
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multi-Part, Single Ascending Dose and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and PK of ATTO1310 in Adult Volunteers, Patients With Atopic Dermatitis, and Patients With Chronic Pruritus
Brief Title: Safety, Tolerability and PK of ATTO-1310 in Healthy Volunteers and Patients With Atopic Dermatitis and Patients With Chronic Pruritus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Attovia Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATTO-1310-101
Record Dates: First submitted 2024-12-26; First posted 2025-01-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Normal Volunteers; Atopic Dermatitis (AD); Atopic Eczema; Chronic Pruritus
Keywords: Atopic dermatitis; AD; Atopic eczema; Eczema; Chronic pruritis; Itch; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Intervention Model Description: Single ascending dose, multiple ascending dose, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ATTO-1310 single dose IV (Experimental): ATTO-1310 Attobody Dose level cohorts receiving a single dose IV
  Interventions: Drug: ATTO-1310
- ATTO-1310 Placebo single dose IV (Placebo Comparator): Placebo preparation to match Experimental Arm with single dose IV
  Interventions: Drug: ATTO-1310 Placebo
- ATTO-1310 single dose SC (Experimental): ATTO-1310 Attobody Dose level cohorts receiving a single dose SC
  Interventions: Drug: ATTO-1310
- ATTO-1310 Placebo single dose SC (Placebo Comparator): Placebo preparation to match Experimental Arm with single dose SC
  Interventions: Drug: ATTO-1310 Placebo
- ATTO-1310 multiple dose SC (Experimental): ATTO-1310 Attobody administered to dose level cohorts in multiple SC doses
  Interventions: Drug: ATTO-1310
- ATTO-1310 Placebo multiple dose SC (Placebo Comparator): Placebo preparation to match Experimental Arm administered in multiple SC doses
  Interventions: Drug: ATTO-1310 Placebo

INTERVENTIONS:
Drug: ATTO-1310 — ATTO-1310 Attobody
  Arms: ATTO-1310 multiple dose SC; ATTO-1310 single dose IV; ATTO-1310 single dose SC
Drug: ATTO-1310 Placebo — Placebo preparation to match ATTO-1310 Dose
  Arms: ATTO-1310 Placebo multiple dose SC; ATTO-1310 Placebo single dose IV; ATTO-1310 Placebo single dose SC

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, and pharmacokinetics of ATTO-1310 in healthy adults, patients with atopic dermatitis and patients with chronic pruritus.

The main questions it aims to answer are:

What medical problems do participants have when taking ATTO-1310? How long does ATTO-1310 stay in the body after dosing? Researchers will compare ATTO-1310 to a placebo (a look-alike substance that contains no drug).

Participants will be dosed with ATTO-1310 or a placebo, visit the clinic for checkups and tests, and keep a diary of their symptoms.

DETAILED DESCRIPTION:
This is a 4-part study. Parts 1 and 2 will be a single and multiple ascending dose design, respectively, assessing the safety, tolerability and PK of ATTO-1310 in healthy adult volunteers. Part 3 and Part 4 will consist of a single dose in adult patients with atopic dermatitis or chronic pruritus, respectively, to assess safety, tolerability, PK, and PD based on biomarkers in the blood.

ELIGIBILITY:
Parts 1 & 2 (Healthy Volunteers) Key Inclusion Criteria:

* Any sex or gender who is 18 to 65 years old
* Body weight of 50 to 125 kg and body mass index (BMI) between 18.5 and 35 kg/m2
* Considered in good general health based on medical history, physical exam, 12-lead ECG, screening clinical laboratory findings, and vital signs
* Negative pregnancy test for subjects of child-bearing potential
* Use of highly effective forms of birth control

Part 3 (Subjects with Atopic Dermatitis) Inclusion Criteria:

* Any sex or gender who is 18 to 65 years old
* Body weight of 50 to 125 kg and BMI between 18.5 and 40 kg/m2
* Clinically confirmed diagnosis of active AD
* At least a 1-year history of AD and had no significant flares in AD for at least 4 weeks before Screening
* Baseline weekly mean of daily PP-NRS ≥ 7 at Day 1
* EASI score of ≥ 7 at Screening and Day 1
* vIGA-AD score of ≥ 3 at Screening and Day 1
* Use of topical bland emollient (moisturizer) once or twice daily for at least 5 of the 7 days immediately before Day 1 and agrees to continue using that same emollient at the same frequency throughout the study
* Negative pregnancy test for subjects of child-bearing potential
* Use of highly effective forms of birth control

Part 4 (Subjects with Chronic Pruritus) Inclusion Criteria:

* Any sex or gender who is 18 to 85 years old
* Body weight of 50 to 125 kg, inclusive, and BMI between 18.5 and 40 kg/m2
* Has had chronic pruritus for at least 6 months and is unresponsive to at least a 2-week course of emollient use.
* Chronic pruritus that affects at least 2 of the following body areas: legs, arms, or trunk
* A single PP-NRS score of ≥ 5 in the 24-hour period prior to the Screening visit
* Baseline weekly mean of daily PP-NRS ≥ 7 at Day 1
* Use of a stable dose of topical bland emollient (moisturizer) once or twice daily for at least 2 weeks before Day 1 and agrees to continue using that same emollient at the same frequency throughout the study
* Negative pregnancy test for subjects of child-bearing potential
* Use of highly effective forms of birth control

Parts 1 & 2 (Healthy Volunteers) Exclusion Criteria:

* Any clinically significant underlying illness.
* History of malignancy within 5 years of Screening, except adequately treated basal carcinoma or in situ carcinoma of the cervix.
* History of major surgery within 8 weeks prior to Day 1
* History of asthma requiring regular use of a bronchodilator or a daily maintenance therapy
* History of hypersensitivity (including anaphylaxis) to a biologic medication, vaccine, an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody), or to any of the IP excipients (sucrose, polysorbate 80, or histidine)
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or is positive for HIV
* Active or latent tuberculosis infection
* Smoking more than 20 cigarettes (or cigars, cigarillos, or e-cigarettes equivalent) per day
* History of drug or alcohol abuse
* Laboratory values outside of the normal range

Exclusion Criteria for Part 3 (Subjects with Atopic Dermatitis):

* Any clinically significant underlying illness
* History of a clearly defined etiology for pruritus other than AD, including but not limited to urticaria, psoriasis, or other non-atopic dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, uncontrolled hyperthyroidism, and infection
* History of malignancy within 5 years of Screening
* History of major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study
* History of asthma requiring regular use of a bronchodilator or a daily maintenance therapy
* History of recurrent eczema herpeticum
* History of known primary immunodeficiency, is considered immunocompromised, history of untreated latent tuberculosis infection, has been treated for active tuberculosis in the past year, or has been treated for a parasitic infection in the past 6 months
* History of major depression
* History of hypersensitivity (including anaphylaxis) to a biologic medication, vaccine, an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody), or to any of the IP excipients (sucrose, polysorbate 80, or histidine)
* Active HBV or HCV or is positive for HIV
* Smoking more than 20 cigarettes (or cigars, cigarillos, or e-cigarettes equivalent) per day
* ECG with a QTcF > 450 msec for males or > 470 msec for females at Screening
* History of drug or alcohol abuse
* Subject has applied topical corticosteroid in the 14 days preceding Day 1
* Subject has used prohibited medications or therapies during the specified washout period before Day 1 (as defined in the protocol)
* Laboratory values outside of the normal range

Exclusion Criteria for Part 4 (Subjects with Chronic Pruritus):

* Primary dermatologic diagnosis associated with pruritic skin lesions at the time of screening
* Regional neuropathic disease associated with pruritus
* Severe renal failure requiring dialysis
* Untreated cholestatic liver disease
* Liver function tests (bilirubin, AST, ALT, alkaline phosphatase) >2.5 times above the upper limit of normal
* History of infectious dermatoses
* Suspected diagnosis of somatoform pruritus
* Suspected diagnosis of drug-induced pruritus
* History of malignancy within 5 years of Screening
* History of unexplained fevers, night sweats, or unintentional weight loss
* Major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study
* History of asthma requiring regular use of a bronchodilator or a daily maintenance therapy
* History of known primary immunodeficiency, is considered immunocompromised, untreated latent tuberculosis infection, has been treated for active tuberculosis in the past year, or has been treated for a parasitic infection in the past 6 months
* History of attempted suicide
* History of hypersensitivity (including anaphylaxis) to a biologic medication, vaccine, an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody), or to any of the IP excipients (sucrose, polysorbate 80, or histidine)
* Active HBV or HCV or is positive for HIV.
* Smoking more than 20 cigarettes (or cigars, cigarillos, or e-cigarettes equivalent) per day
* ECG with a QTcF > 450 msec for males or > 470 msec for females at Screening
* History of drug or alcohol abuse
* Use of prohibited medications as defined in the Protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | 0-113 Days for SAD; 0-143 Days for MAD
  The primary analysis will describe the incidence of AEs and laboratory abnormalities. AEs will be coded according to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA, version 26.1 or the current version). Their severity will be graded using the NCI CTCAE v5.0 or the current version.
Incidence of laboratory abnormalities | 0-113 Days for SAD; 0-143 Days for MAD
  Clinical laboratory parameters (hematologic and blood chemistry) will be summarized for each post-baseline visit.
Incidence of ECG abnormalities | 0-113 Days for SAD; 0-143 Days for MAD
  ECG findings (including QT abnormalities) will be summarized for each post-baseline visit.
Incidence of vital sign abnormalities | 0-113 Days for SAD; 0-143 Days for MAD
  Vital signs (systolic and diastolic blood pressure, temperature, heart rate) will be summarized for each post-baseline visit.

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibodies | 0-113 Days for SAD; 0-143 Days for MAD
  Baseline prevalence of ADA, Changes in ADA status from prior to the first dose of IP to each post-dose timepoint and ADA titer values for samples confirmed positive for ADA will be evaluated to assess the immunogenicity of single and multiple dose levels of ATTO-1310.
Peak plasma concentration (Cmax) ATTO-1310 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include maximum concentration (Cmax)of ATTO-1310
Circulating half-life of ATTO-1310 (t1/2) | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include half-life (t1/2) of ATTO-1310
Area Under the Plasma Concentration Versus Time Curve (AUC) | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include area under the plasma concentration-time curve (AUC).
Clearance rate (C) of ATTO-1310 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include characterization of the Clearance rate (C) of ATTO-1310
Volume of Distribution (V) of ATTO-1310 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include characterization of the Volume of distribution (V) of ATTO-1310
Bioavailability (F) of ATTO-1310 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-1310 in participants will include characterization of the Bioavailability (F) of ATTO-1310

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc.
Locations (15):
- United States (9):
  - Attovia Clinical Site 103, Encinitas, California
  - Attovia Clinical Site 116, Rocklin, California
  - Attovia Clinical Site 107, Sacramento, California
  - Attovia Clinical Site 109, Coral Gables, Florida
  - Attovia Clinical Site 102, Plainfield, Indiana
  - Attovia Clinical Site 104, Saint Joseph, Missouri
  - Attovia Clinical Site 106, Reno, Nevada
  - Attovia Clinical Site 114, New York, New York
  - Attovia Clinical Site 108, San Antonio, Texas
- Canada (6):
  - Attovia Clinical Site 110, Fredericton, New Brunswick
  - Attovia Clinical Site 111, Newmarket, Ontario
  - Attovia Clinical Site 112, Peterborough, Ontario
  - Attovia Clinical Site 113, Toronto, Ontario
  - Attovia Clinical Site 105, Montreal, Quebec
  - Altasciences, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No